CLINICAL TRIAL: NCT00456638
Title: Clinical Study of Depodur Efficacy in Decreasing Post Operative Pain After Off Pump Coronary Artery Bypass Grafting (OP-CABG)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty aquiring investigational drug
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 16402
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2008-04

CONDITIONS: Pain, Postoperative
Keywords: OP-CABG; Depodur traditional drug
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depodur (Experimental): Depodur arm
  Interventions: Drug: Depodur
- Traditional (Active Comparator): traditional management
  Interventions: Drug: Depodur

INTERVENTIONS:
Drug: Depodur — Depodur vs. traditional management
  Other Names: Traditional

SUMMARY:
The purpose of this study is to determine whether epidural Depodur alleviates the pain of OP-CABG surgery. This includes pain associated with sternotomy, retraction, dissection and other tissue insults, as well as the induced inflammatory system and effects from prolonged ventilation in the ICU setting.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether epidural Depodur alleviates the pain of OP-CABG surgery. This includes pain associated with sternotomy, retraction, dissection and other tissue insults, as well as the induced inflammatory system and effects from prolonged ventilation in the ICU setting. It will be compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 18-99 years old
* All patients who will have surgery for OP-CABG

Exclusion Criteria:

* Pregnant females
* Patients with allergy to morphine
* Patients nursing an infant
* Patients with migraine headaches
* Patients taking Coumadin within 7 days or demonstrating INR > 13
* Patients taking Heparin unless documented normal partial thromboplastin time
* Patients taking Clopidogrel in previous 7 days
* Patients taking Ticlopidine in previous 14 days
* Patients taking Aspirin in previous 48 hours
* Patients receiving low molecular weight heparin therapy within 24 hours previous
* Patients with Narcolepsy and/or sleep apnea
* Patients on chronic opioid therapy
* Patients participating in another study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Comparison of pain (Visual Analog Scale), post-op morphine usage, and side effects between the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Jay Horrow, MD, Study Chair — Drexel University College of Medicine